CLINICAL TRIAL: NCT07073014
Title: A Phase 3, Open-Label, Long-Term Extension Study to Evaluate the Safety and Efficacy of Vosoritide in Children With Hypochondroplasia
Brief Title: Long-Term Extension Study of Vosoritide to Treat Children With Hypochondroplasia
Acronym: CANOPY-HCH-EXT
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111-308
Record Dates: First submitted 2025-06-27; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hypochondroplasia
MeSH Terms: conditions — Hypochondroplasia | interventions — vosoritide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vosoritide (Experimental): Open-label active drug
  Interventions: Drug: Vosoritide

INTERVENTIONS:
Drug: Vosoritide — Open-label administration of vosoritide using weight-band dosing

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of daily doses of vosoritide in participants with HCH

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed the Week 52 visit for 111-303 or 111-212 and have open epiphyses as assessed by left hand antero-posterior (AP) X-rays
* Parent(s) or guardian(s) must be willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to performance of any study-related procedure
* Females ≥ 10 years old or who have begun menses must have a negative pregnancy test at the Baseline visit and be willing to have additional pregnancy tests during the study
* If sexually active, participants must be willing to use a highly effective method of contraception while participating in the study
* Participants are willing and able to perform all study procedures as physically possible
* Parent(s) or caregiver(s) are willing to administer daily injections to the participants and willing to complete the required training

Exclusion Criteria:

* Permanently discontinued study treatment in the studies 111-303 or 111-212
* Evidence of decreased growth velocity (AGV < 1.5 cm/year) as assessed over a period of at least 6 months and growth plate closure assessed as per standard of care
* Taking or planning to take any prohibited medications
* Planned or expected to have limb-lengthening surgery during the study period
* Planned or expected bone-related surgery during the study period
* Require any investigational agent prior to completion of study period
* Have current malignancy, history of malignancy, or currently under work-up for suspected malignancy
* Have known hypersensitivity to vosoritide or its excipients
* Is pregnant or breastfeeding at Baseline or planning to become pregnant (self or partner) at any time during the study
* Concurrent disease or condition that, in the view of the investigator, would interfere with study participation or safety evaluations, for any reason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the long-term efficacy of vosoritide treatment until final adult height (FAH) | Annually from enrollment through Final Adult Height, defined as 16 years of age for females and 18 years of age for males
  As measured by change from baseline in height Z-score

SECONDARY OUTCOMES:
Evaluate the maintenance effect of vosoritide treatment on standing height | Baseline to week 52
  change from baseline in height at Week 52
Evaluate the maintenance effect of vosoritide treatment on standing height Z-score | Baseline to week 52
  Change from baseline in height Z-score at Week 52
Evaluate long-term effect of vosoritide treatment on growth velocity | Annually from enrollment through Final Adult Height, defined as 16 years of age for females and 18 years of age for males
  Absolute 6- or 12-month interval AGV
Evaluate long-term effect of vosoritide treatment on body proportionality | Annually from enrollment through Final Adult Height, defined as 16 years of age for females and 18 years of age for males
  Change from baseline in upper to lower body segment ratio
Evaluate long-term effect of vosoritide treatment on bone age versus chronological age | Annually from enrollment through Final Adult Height, defined as 16 years of age for females and 18 years of age for males
  As measured by left-hand and wrist x-ray
Evaluate long-term effect of vosoritide treatment on bone metabolism biomarkers | Annually from enrollment through Final Adult Height, defined as 16 years of age for females and 18 years of age for males
  Change from baseline in serum collagen X marker
Evaluate long-term changes in Health-Related Quality of Life (HRQoL) | Annually from enrollment through Final Adult Height, defined as 16 years of age for females and 18 years of age for males
  Change from baseline as measured by Quality of Life In Short-Statured Youth (QoLISSY) total score
Evaluate long-term effect of vosoritide treatment on bone quality | Annually from enrollment through Final Adult Height, defined as 16 years of age for females and 18 years of age for males
  Change from baseline in bone mineral density (BMD) as measured by Dual X-Ray Absorptiometry
Evaluate long-term effect of vosoritide treatment on pubertal growth as measured by Tanner Staging | Annually from enrollment through Final Adult Height, defined as 16 years of age for females and 18 years of age for males
To monitor the incidence of otitis media | Annually from enrollment through Final Adult Height, defined as 16 years of age for females and 18 years of age for males
To monitor the frequency of seizures | Annually from enrollment through Final Adult Height, defined as 16 years of age for females and 18 years of age for males

CONTACTS AND LOCATIONS:
Locations (23):
- United States (4):
  - Nemours Children's Hospital, Delaware (Alfred I. Dupont Hospital for Children), Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- Canada (3):
  - University of Alberta Stollery Children's Hospital, Edmonton, Alberta
  - SickKids - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- France (4):
  - Hospices Civils de Lyon - Hopital Femme Mere Enfant, Lyon
  - Hopital de la Timone, Marseille
  - Hopital Necker-Enfants Malade, Paris
  - CHU de Toulouse, Toulouse
- Germany (2):
  - Uniklinik Koln, Cologne
  - Univeristatskinderklinik Magdeburg, Magdeburg
- Italy (3):
  - Instituto Giannina Gaslini, Genoa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Ospedale Pediatrico Bambino Gesu, Rome
- Japan (4):
  - Osaka University Hosptial, Osaka
  - Tokushima University Hospital, Tokushima
  - Institute of Science Tokyo Hospital, Tokyo
  - Tottori University Hospital, Tottori
- Vithas Hospital San Jose, Vitoria-Gasteiz, Spain
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided